CLINICAL TRIAL: NCT00966264
Title: Hysterectomy and Levonorgestrel-releasing IUS in the Treatment of Menorrhagia
Brief Title: Hysterectomy and Levonorgestrel Releasing Intrauterine System (LNG-IUS) in the Treatment of Menorrhagia
Acronym: VUOKKO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Eastern Finland (Other); University of Oulu (Other); Tampere University (Other); University of Turku (Other)
Responsible Party: Ritva Hurskainen, project manager, Helsinki University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Finnish Academy-project 29168
Record Dates: First submitted 2009-01-20; First posted 2009-08-26 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Menorrhagia
Keywords: randomized controlled trial; menorrhagia; LNG-IUS; hysterectomy
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNG-IUS (Active Comparator): Levonorgestrel releasing intrauterine system
  Interventions: Drug: LNG-IUS; Procedure: Hysterectomy
- Hysterectomy (Other): Hysterectomy
  Interventions: Drug: LNG-IUS; Procedure: Hysterectomy

INTERVENTIONS:
Drug: LNG-IUS — LNG-IUS releasing 25 microg of levonorgestrel
  Other Names: Mirena
Procedure: Hysterectomy — operation
  Other Names: Removal of uterus by laparoscopy, vaginally or abdominally

SUMMARY:
A randomised study including 236 women referred for essential menorrhagia to five university hospitals in Finland was conducted to compare the cost-effectiveness and the quality of life issues in the treatment of menorrhagia.Participants were randomly assigned to treatment with LNG-IUS (n=119), or hysterectomy (n=117), and were monitored for ten years. The primary outcome measures were health related quality of life (HRQoL), other measures of psychosocial well-being (anxiety, depression, sexual functioning), and costs.

DETAILED DESCRIPTION:
A randomized VUOKKO trial was conducted between 1994-2008 to study hysterectomy and LNG-IUS in the treatment of menorrhagia.Overall, 236 women aged 35 to 49 years who were menstruating, had completed their family size, and were eligible for both treatments were randomized to either receive a LNG-IUS (n=119) or undergo hysterectomy (n=117). The follow-up visits took place six months and 12 months after the treatment, and again five and ten years after the randomization. The primary outcome measures were health related quality of life (HRQoL), other measures of psychosocial well-being (anxiety, depression, sexual functioning), and costs. The amount of menstrual blood loss was objectively measured before treatment and after one and five years. The one year the results were published in 2001 (Lancet 2001;357:273) and the five year results in 2004 (JAMA 2004; 291:1456).

ELIGIBILITY:
Inclusion Criteria:

* heavy menstrual bleeding
* 35-49 years
* were menstruating
* had completed their family size
* were eligible for both treatments

Exclusion Criteria:

* submucous fibroids
* endometrial polyps
* ovarian tumours or cysts,
* cervical pathology
* urinary and bowel symptoms or pain due to large fibroids
* lack of indication for hysterectomy
* history of malignancies
* menopause
* severe depression
* metrorrhagia as a main complaint
* previous treatment failure with LNG-IUS
* severe acne
* uterine malformation

Ages: 35 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 1994-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritva S Hurskainen, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Jorma Paavonen, prof, Study Director — University of Helsinki; Juha Teperi, prof, Study Chair — National Istitute For Health and Welfare, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred and thirty-six women referred for essential menorrhagia to five university hospitals in Finland were randomly assigned to treatment with LNG-IUS (n= 119) or hysterectomy (n=117).
Pre-assignment Details: All randomised women were analysed as intention-to-treat
Groups:
- LNG-IUS: Levonorgestrel releasing intrauterine system (LNG-IUS)
- Hysterectomy: Hysterectomy (abdominal,laparoscopical or vaginal)
Period: Overall Study
Arm/Group | LNG-IUS | Hysterectomy
Started | 119 | 117
Completed | 115 (5 years results) | 114 (5 years results)
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG-IUS | Hysterectomy | Total
Number analyzed (Participants) | 119 | 117 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 117 | 236
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (3.5) | 43.0 (3.2) | 43 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 117 | 236
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: HRQoL (Health Related Quality of Life)
Description: HRQoL was measured by the 5-Dimensional EuroQol (EQ-5D) questionnaire which measures HRQoL in 5 dimensions of life (scale 0-1)(from very poor=0 to very good=5). The results are the change of HRQoL from baseline at 5 years (EQ-5D score at 5 years - EQ-5D score at baseline)
Time Frame: baseline and 5 years
Population: The power calculation was made on the basis of an EQ-5D score SD of 19% and alfa=0.05. The study had 80% power to detect a 7.5% difference between the groups
Measure: Mean (95% Confidence Interval); unit: points on a scale
Arm/Group | LNG-IUS | Hysterectomy
Number analyzed (Participants) | 115 | 114
points on a scale | 0.08 [0.03 to 0.13] | 0.10 [0.05 to 0.15]

2. Primary Outcome: Costs
Time Frame: baseline, 6 and 12 months, 5 and 10 years
Reporting Status: Not Posted, anticipated posting 2010-05
Measure: Number

3. Secondary Outcome: Depression
Time Frame: baseline, 6 and 12 months, 5 and 10 years
Reporting Status: Not Posted, anticipated posting 2010-05

ADVERSE EVENTS:
Arm/Group | LNG-IUS | Hysterectomy
Serious Adverse Events (participants affected / at risk) | 0 | 5
Other Adverse Events (participants affected / at risk) | 80 | 25
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | LNG-IUS | Hysterectomy
bladder perforation (Surgical and medical procedures) | 0/50 (0) | 3/109 (3)
peritonitis (Surgical and medical procedures) | 0/50 (0) | 1/109 (1)
vesicovaginal fistula (Surgical and medical procedures) | 0/50 (0) | 1/109 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 20% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | LNG-IUS | Hysterectomy
hormonal symptoms (Surgical and medical procedures) | 18/119 (18) | 0/117 (0)
menstrual bleeding problems (Surgical and medical procedures) | 61/119 (61) | 2/117 (2)
wund infection (Surgical and medical procedures) | 9/50 (9) | 20/109 (20)
perioperative bleeding (Surgical and medical procedures) | 1/50 (1) | 1/109 (1)
postoperative bleeding (Surgical and medical procedures) | 1/50 (1) | 2/109 (2)
urinary retention (Surgical and medical procedures) | 1/119 (1) | 4/117 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes